CLINICAL TRIAL: NCT03716388
Title: Fecal Microbiota Therapy Vs 5-aminosalicylates for Induction of Remission in Newly Diagnosed Mild-moderately Active UC : a Pilot Study
Brief Title: Fecal Microbiota Therapy Vs 5-aminosalicylates for Induction of Remission in Newly Diagnosed Mild-moderately Active UC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dayanand Medical College and Hospital (Other)
Collaborators: Colitis & Crohn's Foundation (India) (Unknown)
Responsible Party: Principal Investigator, Ajit Sood, Professor and Head, Gastroenterology, Dayanand Medical College and Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-362
Record Dates: First submitted 2018-10-21; First posted 2018-10-23 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Ulcerative Colitis Chronic Mild; Ulcerative Colitis Chronic Moderate
Keywords: Fecal Microbiota Transplantation; Ulcerative Colitis; Induction of Remission
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Fecal Microbiota Transplantation; Mesalamine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FMT Vs Placebo (Experimental): Fecal microbiota transplantation (fresh sample, colonoscopic administration at weeks 0,2,6,10,14) plus placebo granules (4g/day)
  Interventions: Biological: Fecal Microbiota Transplantation; Other: Placebo granules
- FMT Vs Mesalamine (Active Comparator): Fecal microbiota transplantation (fresh sample, colonoscopic administration at weeks 0,2,6,10,14) plus mesalamine granules (4g/day)
  Interventions: Biological: Fecal Microbiota Transplantation; Drug: Mesalamine Granules
- Placebo Infusion Vs Mesalamine (Active Comparator): Placebo infusion (colonoscopic administration at weeks 0,2,6,10,14) plus mesalamine granules (4g/day)
  Interventions: Drug: Mesalamine Granules; Other: Placebo infusion

INTERVENTIONS:
Biological: Fecal Microbiota Transplantation — Freshly passed stools (80 g) will be diluted with normal saline (200 ml) and homogenized using a blender, filtered, filled into 4 syringes (50 ml each) and used within 1 hour of preparation or 6 hours of passage of stools. Polyethylene glycol lavage will be done for bowel preparation and the slurry administered into the ileum and/or caecum by colonoscopy. Post FMT, recipients will be encouraged to retain the slurry for 4-6 hours. FMT sessions will be scheduled at weeks 0,2,6,10,14.
  Arms: FMT Vs Mesalamine; FMT Vs Placebo
Drug: Mesalamine Granules — Mesalamine granules 4 grams a day
  Other Names: Rowasa
  Arms: FMT Vs Mesalamine; Placebo Infusion Vs Mesalamine
Other: Placebo infusion — Water with food grade colour to resemble fecal slurry
  Arms: Placebo Infusion Vs Mesalamine
Other: Placebo granules — Granules resembling mesalamine granules, 4 grams a day
  Arms: FMT Vs Placebo

SUMMARY:
Ulcerative colitis is a chronic idiopathic inflammatory disease of the colon that is characterized by abdominal pain and bloody diarrhea. The pathogenesis of UC involves a complex interplay of genetic factors, immune dysregulation and environmental triggers. Conventional therapies for UC (including 5-aminosalicylates, corticosteroids, azathioprine or 6-mercaptopurine and biologics) focus on altering the immune response by suppression of immune cells. However, the primary pathogenic mechanism underlying UC maybe gut microbiota dysbiosis and a dysfunctional intestinal barrier resulting in an aberrant host immune response. Several studies have shown reduced microbial diversity in UC patients with under representation of anti-inflammatory phyla (Bacteroides and Firmicutes), and a relative increase of pro-inflammatory phyla (Proteobacteria and Actinobacteria). Motivated by this, therapies targeting intestinal dysbiosis (prebiotics, probiotics, synbiotics and fecal microbiota transplant (FMT)) have thus been tried in patients with UC. Though several case series and subsequently four high quality randomized controlled trails have established the efficacy of FMT in induction of remission in active UC, all these studies have used it as an add-on therapy, along with the previously ongoing conventional therapies. The investigators aim to assess the safety and efficacy of FMT as the sole modality for induction of remission in patients with newly diagnosed active UC.

DETAILED DESCRIPTION:
This will be a prospective randomised placebo-controlled trial. Newly diagnosed treatment naive patients with mild to moderately severe UC will be recruited (n=15). The patients will be randomized into 3 groups; i.e group I (n=5): FMT with placebo, group II (n=5): FMT with mesalamine, group III (n=5): Placebo infusion with mesalamine. The patients will undergo colonoscopic administration of fecal slurry (groups I and II) or placebo (group III) at weeks 0,2,6,10 and 14. Mesalamine will be administered in a dose of 4g/day. In case of clinical worsening during the study, a short course of steroids will be added. The primary end point will be clinical remission (Mayo score ≤2, all subscores ≤ 1) at week 14. Secondary end points will be achievement of endoscopic remission (endoscopic Mayo score 0) and histological remission (Nancy grade 0, 1) at the end of 14 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Active UC:

  1. UC diagnosed based on history of chronic (>4 weeks), inflammatory (with blood and mucous) diarrhoea
  2. Total Mayo Score 4-10, Mayo endoscopic sub-score of >1
  3. Histopathology suggestive of UC

Exclusion Criteria:

* Severe UC (Total Mayo 11-12, Endoscopic Mayo Score 3)
* Uncertainty about diagnosis of UC : Infective colitis/ Indeterminate Colitis/ Crohn's Colitis
* Associated irritable bowel syndrome (IBS)
* Past history of surgery or colorectal surgery
* Exposure to antibiotics or probiotics in the last 4 weeks
* Patients with evidence of infections like C. difficile, cytomegalovirus, HIV, parasitic infections or extra-intestinal infections requiring antibiotics.
* Significant cardiopulmonary co-morbidities (high risk for repeated colonoscopy)
* Pregnancy
* Refusal to consent for repeated colonoscopies.

Donor

* Single donor (voluntary healthy individual) after informed consent
* Inclusion criteria for donor

  * No personal or family history of UC or any other autoimmune disease or malignancy
  * Screened by stool microscopy and culture for common detectable enteric pathogens (Salmonella, Shigella, Campylobacter, Vibrio cholera, E. coli, Clostridium difficile, Giardia lamblia and Cryptosporidium) at the start of the study and every 4 weeks thereafter.
  * Negative for antibodies against hepatitis A, C and E, hepatitis B surface antigen (HBsAg), syphilis and human immunodeficiency virus (HIV).
* Exclusion criteria for donor

  * High-risk sexual behaviors
  * Communicable illnesses
  * Antibiotic treatment within the past 3 months
  * Intrinsic gastrointestinal illnesses such as irritable bowel syndrome, inflammatory bowel disease, gastrointestinal malignancies or major gastrointestinal surgical procedures
  * Ongoing immune-modulator therapy for any concurrent illness
  * Chronic pain syndromes
  * Neurologic/neurodevelopmental disorders
  * Metabolic syndrome
  * Obesity (BMI >30 kg/m2)
  * Malignant illnesses
* Donor's diet will be monitored with a diet diary.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Clinical remission | Week 14
  Mayo score ≤2, each subscore ≤1

SECONDARY OUTCOMES:
Clinical response | Weeks 0,2,6,10,14
  Reduction of Mayo score ≥30% and ≥3 points compared to baseline
Endoscopic remission | Week 14
  Endoscopic Mayo subscore 0
Histological remission | Week 14
  Nancy grade 0 or 1

CONTACTS AND LOCATIONS:
Overall Officials: Ajit Sood, DM, Principal Investigator — Professor and Head Gastroenterology
Locations (1):
- Dayanand Medical College and Hospital, Ludhiana, Punjab, India

IPD SHARING:
Plan to Share IPD: Undecided